CLINICAL TRIAL: NCT06874530
Title: Efficacy of Isatuximab-basedregimens in Relapsed/Refractory Multiple Myeloma With 1q21+
Brief Title: Efficacy of Isatuximab-based Regimens in Relapsed/Refractory Multiple Myeloma With 1q21+
Acronym: Isa_1q21+
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: Isa_1q21+
Record Dates: First submitted 2024-12-03; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-11

CONDITIONS: Multiple Mieloma
Keywords: Relapsed; Refractory; Isatuximab; 1q21+
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Analysis group that based on cytogenetic profile has 1q21 aberrations.: Analysis group that based on cytogenetic profile has 1q21 aberrations.
- Analysis group that based on cytogenetic profile absent for 1q21 aberration.: Analysis group that based on cytogenetic profile absent for 1q21 aberration.

SUMMARY:
This is a non-interventional, national, multicentre retrospective and prospective observational study aiming at assessing the efficacy of isatuximab-based regimens in RRMM patients with 1q21+ in a real-life setting.

Due to the limited information as to isatuximab's impact in real-world settings and that MM is a rare cancer, patients will be enrolled both prospectively and retrospectively from approximately 8 haematologic/oncologic centers in Italy. Prospective enrollment will allow an assessment of true baseline and the beneficial treatment of isatuximab among RRMM patients with 1q21+. The inclusion of retrospectively enrolled patients previously exposed to isatuximab-based regimens (Isa-Pd and Isa-Kd) will allow for maximal data capture to evaluate isatuximab treatment as part of routine care.

All the sites participating in the study are using isatuximab-based regimens for the treatment of RRMM patients in clinical practice. According to data availability and/or clinical experience of the sites, data from approximately 150 patients consecutively treated in the participating centers will be collected in the present study and compared with data published in the literature.

DETAILED DESCRIPTION:
This is a non-interventional, national, multicentre retrospective and prospective observational study aiming at assessing the efficacy of isatuximab-based regimens in RRMM patients with 1q21+ in a real-life setting.

Due to the limited information as to isatuximab's impact in real-world settings and that MM is a rare cancer, patients will be enrolled both prospectively and retrospectively from approximately 8 haematologic/oncologic centers in Italy. Prospective enrollment will allow an assessment of true baseline and the beneficial treatment of isatuximab among RRMM patients with 1q21+. The inclusion of retrospectively enrolled patients previously exposed to isatuximab-based regimens (Isa-Pd and Isa-Kd) will allow for maximal data capture to evaluate isatuximab treatment as part of routine care.

All the sites participating in the study are using isatuximab-based regimens for the treatment of RRMM patients in clinical practice. According to data availability and/or clinical experience of the sites, data from approximately 150 patients consecutively treated in the participating centers will be collected in the present study and compared with data published in the literature.

Patients will receive or will have been previously prescribed isatuximab in combination with either pomalidomide and dexamethasone (Isa-Pd) or carfilzomib and dexamethasone (Isa-Kd), in routine clinical practice and independently of the proposal to be enrolled into this study.Given the observational nature of the study, the decision of the patients to take part in this study will have no impact on the current and/or future care they receive and patient current therapy, if any, will be maintained with no change.

No clinical study visits are mandated; visits will be scheduled by the treating physician according to patients-specific needs and local standard of care (SoC).

After receiving the signed informed consent form from the patient, the investigator will start documenting retrospective and prospective data using electronic data capture. Each investigator should collect data from patients fulfilling all inclusion and exclusion criteria. After confirmation of the patient'seligibility, the patient's last visit, baseline characteristics, MM-related data and therapy-related data will be documented in the Case Report Form.

The primary objective of this retrospective and prospective study is to evaluate the efficacy of isatuximab-based regimens (Isa-Pd and Isa-Kd) for RRMM with 1q21+ in a real-life setting.

Secondary objectives aim at: • exploring the safety and tolerability profile of isatuximab-based regimens in RRMM patients with or without 1q21+ • defining which clinical and cytogenetic risk factors may be associated with 1q21+ (both gain and amplification) • exploring the prognostic impact of different 1q21+ subtypes (gain and amplification) in patients with RRMM, in terms of efficacy, safety and tolerability.

Two groups of analysis will be identified according to the cytogenetic profile (presence or absence of 1q aberrations). The efficacy of isatuximab-based regimens Isa-Pd and Isa-Kd in real-world practice will be compared among RRMM patients with and without 1q21 alteration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signed Informed Consent form (whenever feasible)
* Diagnosis of RRMM prior exposed to >1 lines of therapies including Isatuximab-based regimens
* Availability of FISH results, including 1q2, at diagnosis and/or at relapse

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study participants will be adult patients with a diagnosis of RRMM with chromosomal 1q21 abnormality, previously exposed to >1 lines of therapies including isatuximab-based regimens outside clinical trials.
  The study will aim to enroll up to approximately 150 patients with a recorded diagnosis of RRMM 1q21+, from various Italian clinical sites.
  All eligible patients will be consecutively proposed to be enrolled in the study. Patients will be asked to take part to the present study in the context of a follow-up visit, as per standard care practice. Documentation that informed consent occurred prior to the subject's entry into the study should be recorded in the subject's source documents.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Hematologic response rate, according to the International Myeloma Working Group (IMWG) criteria8 in RRMM with 1q21+ treated with Isa-PD and Isa-KD | Within 12 months from the beginning of therapy.
  The proportion of patients with stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response (PR) as best overall response assessed by Investigator using the IMWG response criteria.

SECONDARY OUTCOMES:
PFS in RRMM with 1q21+ treated with Isa-Pd and Isa-Kd | 12 months after therapy initiation
  Time from isatuximab start date to the date of first documentation of progressive disease (PD), as determined by the Investigator, or the date of death from any cause, whichever comes first.
TTP in RRMM with 1q21+ treated with Isa-PD and Isa-KD | 12 months from the start of treatment.
  Time from the initiation of isatuximab until progressive the according to the Common Terminology Criteria for Adverse Events v5.0 (CTCAE)
Cytogenetic profile in RRMM patients with 1q21+. | Baseline
  Evaluation by FISH analysis
Minimal residual disease (MRD) in patients with and without 1q21+ treated with isatuximab | perioperatively/periprocedurally
  MRD negativity and sustained MRD negativity in patients with at least VGPR, sCR, or CR to determine the depth of response at the molecular level, where data are available as per standard of care.
  The MRD will be measured by next-generation sequencing in bone marrow aspiration whena vailable (sensitivity of 10-5).
MRD in RRMM with gain(1q21) or amp(1q21) treated with isatuximab-based regimens. | through study completion, once a year, an avarage of 2 years
  Difference in the outcomes of patients with gain(1q21) and amp(1q21) treated with Isa-Pd/Isa-Kd.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Azienda Ospedaliera-Universitaria di Bologna, Bologna, Italy